CLINICAL TRIAL: NCT01898468
Title: Post-Thoracotomy Pain Syndrome: A Randomized, Double Blind, Study Comparing Closure Techniques
Brief Title: Post-Thoracotomy Closure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHN13-5894
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2018-10

CONDITIONS: Post Thoracotomy Pain Syndrome
Keywords: Neuropathic pain symptoms; Intracostal Closure Technique; Pericostal Suture Closure Technique; Post surgical pain; Post thoracotomy pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracostal Closure Technique (Active Comparator): Closure involves drilling four evenly spaced holes using a 5-mm bit attached to the end of a Stryker drill into the bed of the sixth rib.
  Interventions: Procedure: Intracostal Closure Technique
- Pericostal Closure Technique (Active Comparator): Closure involves placing sutures around the ribs in the standard pericostal fashion
  Interventions: Procedure: Pericostal Closure Technique

INTERVENTIONS:
Procedure: Pericostal Closure Technique
  Arms: Pericostal Closure Technique
Procedure: Intracostal Closure Technique
  Arms: Intracostal Closure Technique

SUMMARY:
Post-thoracotomy Pain Syndrome (PTPS) is defined as "pain that recurs or persists along a thoracotomy scar at least 2 months following surgery." PTPS presents a frustrating challenge to patients and healthcare providers alike. PTPS can affect up to 80% of patients undergoing thoracotomies, and results in significant impairment. A proposed mechanism for PTPS is the compression of the intercostal nerves during routine closure. Closure of thoracotomies using intracostal sutures is a novel technique where sutures are passed through holes drilled into the rib; thus, avoiding compression of the nerves. We propose a double-blind, randomized control study involving 90 patients undergoing elective posterolateral thoracotomies. Participants will be randomly assigned to undergo thoracotomy closure with pericostal sutures or intracostal sutures. Our primary outcome will assess the incidence and severity of PTPS at 3, 6, and 12 months after surgery between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-88 years age
* Patients undergoing surgery with an open thoracotomy incision

Exclusion Criteria:

* Patient refusal
* Inability to give informed consent
* Concurrent drug addiction or methadone use
* Present chronic pain syndrome
* Significant psychiatric illness excluding depression
* Cannot understand English, read or write in English independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of post-thoracotomy pain | 3 months post surgery
  A Numerical Rating Score (NRS) for maximal daily pain from the patients surgical incision will also be measured (0 = no pain, 10 = worst possible pain) 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (2):
- Canada (2):
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario